CLINICAL TRIAL: NCT04959708
Title: Online Physical Therapy Management for Physiotherapists to Cope Psychological Distress During Covid-19 Pandemic
Acronym: PHYSFORPHYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Cristina Bravo, Dr, Universitat de Lleida
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHYSFORPHYS
Record Dates: First submitted 2021-07-07; First posted 2021-07-13 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Psychological Distress
Keywords: physical therapy; Covid-19; anxiety; depression; body awareness
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: A clinical pilot study will be conducted with two controlled and parallel groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants and the therapist will remain unblinded, however, the rest of group researcher will be blinded during the whole study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participants in the control group will have the same exposure in time as the intervention group and will be asked to maintain their lifestyle during the whole study and to refrain from starting any new regular physical activity. In case they can not maintain the same lifestyle during the study period, they will be asked to inform the researchers at any of the assessments.
  Interventions: Other: Insula treatment
- Intervention group (Experimental): The intervention group will consist of the Ínsula method. Insula method will be developed twice a week for 12 weeks online form through videoconference platform. The intervention will consist of twelve individual treatments. Insula method consists of the facilitation and activation of self-regulation resources, relational regulation through breathing, movement, contact, sensory stimulation and posture
  Interventions: Other: Insula treatment

INTERVENTIONS:
Other: Insula treatment — he intervention will consist of twelve individual treatments. Insula method consists of the facilitation and activation of self-regulation resources, relational regulation through breathing, movement, contact, sensory stimulation and posture

SUMMARY:
This project is aimed at physiotherapists and physiotherapy students who have been psychologically affected during the COVID 19 pandemic.

The objective of the approach is to generate a free intervention programme in virtual modality, from the approach of physiotherapy in mental health, which would help them to alleviate the negative effects of the pandemic, offer them coping tools and collaborate to improve their state of well-being.

DETAILED DESCRIPTION:
The intervention group will consist of the Ínsula method. Insula method will be developed twice a week for 12 weeks online form through videoconference platform. The intervention will consist of twelve individual treatments. It is a program of Physiotherapy in Mental Health, created by the physiotherapists Eugenia de León (Guatemala) and Moisés Magos (Mexico) in conjunction with the Psychiatrist Roberto Martínez Porras (Guatemala). It has a progressive design, seeking to strengthen emotional self-regulation skills, connection with others and the environment, and to guide a self - knowledge process. All these objectives are worked through body resources, like conscious movement, breathing, posture, contact, relaxation exercises, etc. The program has influence of various other disciplines such as Tai - Chi, Chi Kung, Sensorimotor Therapy, Somatic Education, Mindfulness, BBAT, among others. Likewise, its principles and progression are based on theoretical models of Neurosciences

ELIGIBILITY:
Inclusion Criteria:

* they are physiotherapist with a moderate or severe psychological distress self-perceived regarding COVID-19 pandemic
* age >18 years
* they can manage to stand from the position of "lying", "sitting", and "standing" without assistance
* they can have smartphone, laptop or device and internet access to follow the intervention

Exclusion Criteria:

* they could not follow the intervention due to cognitive or physical health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Scale Body Connection | Baseline and up to 12 weeks and 1 year
  The scale consists of 20 items scored on a Likert scale ranging from 0 ("not at all") to 4 ("all the time"). It includes two independent factors (r=-.08). The first factor is Body Awareness, which assesses conscious attention to sensory cues that indicate the state of the body (e.g., tension, nervousness, relaxation). The second factor, bodily dissociation, measures bodily connection to or detachment from emotional experiences. The internal consistency of both factors was considered suitable on the basis of a Cronbach's α of 0.83 for BA (12 items) and 0.78 for BD (8 items)

SECONDARY OUTCOMES:
Depression anxiety and stress scale | Baseline and up to 12 weeks and 1 year
  This questionnaire clearly differentiates anxiety from depression. Patients rate the frequency and severity of 21 negative emotional symptoms they have experienced during the previous week, using a scale ranging from 0 to 3. The questionnaire consists of three scales (depression, anxiety and stress) containing 7 items each. It is a questionnaire that allows a brief assessment of the three most important aspects of minor psychiatric disorders: depression, anxiety and stress
Warwick-Edinburgh Mental Well-being Scale | Baseline and up to 12 weeks and 1 year
  It measures mental well-being in the previous two weeks. It is an ordinal scale consisting of 14 items with positive statements. Each item offers a 5-point Likert-type scale, from "Not at all" to "All the time", and an overall score is obtained by summing all items (range 14-70); higher scores indicate higher levels of mental well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Cristina Bravo Navarro, Igualada, Barcelona, Spain